CLINICAL TRIAL: NCT04542005
Title: Cost Effectiveness Analysis of a Randomized Control Trial of q3h vs. q4h Albuterol as Discharge Criteria From the Hospital for Pediatric Asthma Exacerbations
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not obtained
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Raymond Parlar-Chun, Assistant Professor of Pediatrics, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HSC-MS-20-0604
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Asthma in Children
Keywords: albuterol; asthma exacerbation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- q3h albuterol (Experimental): Using q3h as discharge criteria from hospital
  Interventions: Behavioral: q3h albuterol
- q4h albuterol (No Intervention): Using q4h as discharge criteria from hospital

INTERVENTIONS:
Behavioral: q3h albuterol — Using q3h albuterol as discharge criteria from hospital
  Arms: q3h albuterol

SUMMARY:
Asthma is the most common chronic condition among children, and the third leading reason for hospitalization of children in the United States. It exerts a large healthcare burden on the US with estimated annual direct healthcare cost of approximately $50.1 billion with indirect costs of $5.9 billion.

Asthma is characterized by airway inflammation and airway constriction. Albuterol and other betaagonists are first line standard of care for acute exacerbations and provide short acting smooth muscle relaxation and subsequent airway opening. The frequency of albuterol administration is dependent on the severity of the exacerbation. For hospitalized patients here at Children's Memorial Hermann (CMHH), patients may receive nebulized albuterol continuously or if the exacerbation is not as severe, receive albuterol intermittently. Intermittent albuterol frequency ranges from every two hour treatments, every three hour (q3h) treatments, or every four hour (q4h) treatments. As patients recover from their acute exacerbation, their frequency of albuterol administration is progressively titrated along this continuum. Expert consensus uses q4h albuterol as discharge criteria from the hospital. However, recent QI initiatives have studied the effect of q3h treatments as the discharge cutoff with no reported changes in safety or harm. There are no randomized controlled trials available. Furthermore, there are no economic evaluations available to see if costs saved by decreasing the length of hospital care are merely being shifted to subsequent clinic or emergency room care costs.

The investigators aim to conduct a randomized control trial to compare q3h vs. q4h albuterol as hospital discharge criteria for patients admitted for acute asthma exacerbations. The investigators also propose to conduct a costeffectiveness analysis of the trial. If the hypothesis that q3h albuterol is safe and as effective as q4h albuterol as discharge criteria, the investigators would be able to argue for a new standard of care that is more cost effective for this very costly and common disease of children in the United States

ELIGIBILITY:
Inclusion Criteria:

* Children with Primary Reason for Hospitalization of Asthma Exacerbation

Exclusion Criteria:

* Those that never needed q3h albuterol treatments

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Total Treatment Days | Hospitalization to 15 days after discharge

SECONDARY OUTCOMES:
Total Costs | Hospitalization to 15 days after discharge

IPD SHARING:
Plan to Share IPD: Undecided